CLINICAL TRIAL: NCT03577730
Title: Caffeine and Neurologic Recovery Following Surgery and General Anesthesia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Phillip Vlisides, Assistant Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00135919
Record Dates: First submitted 2018-06-08; First posted 2018-07-05 (Actual); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Pain, Postoperative
Keywords: Opioid Use; Opioid Dependence; Opioid-Related Disorders; Opioid Abuse; Opioid-use Disorder; Pain; Pain, Postoperative; Cognitive Impairment; Delirium; Delirium on Emergence; Depression; Anxiety; Anxiety Disorders; Affect
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders; Pain; Cognitive Dysfunction; Delirium; Emergence Delirium; Depression; Anxiety Disorders | interventions — caffeine citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a single-center, quadruple-blinded, pilot randomized controlled trial at the University of Michigan Health System.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Prepared intravenous piggyback solution of caffeine citrate (200 mg caffeine) will be directly delivered to the operating room prior to the surgery of enrolled participants who are randomized to this group.
  Interventions: Drug: Caffeine Citrate
- Control (Placebo Comparator): Prepared intravenous piggyback solution of 5 percent dextrose water will be directly delivered to the operating room prior to the surgery of enrolled participants who are randomized to this group.
  Interventions: Drug: Dextrose Water

INTERVENTIONS:
Drug: Caffeine Citrate — Prepared intravenous piggyback solutions of caffeine citrate (200 mg caffeine) will be directly delivered to the operating room prior to the surgery of enrolled participants.
  Arms: Experimental
Drug: Dextrose Water — Prepared intravenous piggyback solutions of 5 percent dextrose water will be directly delivered to the operating room prior to the surgery of enrolled participants.
  Arms: Control

SUMMARY:
The ongoing opioid epidemic is a public health crisis, and surgical patients are particularly vulnerable to opioid-dependency and related risks. Emerging data suggest that caffeine may reduce pain after surgery. Thus, the purpose of this study is to test whether caffeine reduces pain and opioid requirements after surgery. The investigators will also test whether caffeine improves mood and brain function (e.g., learning, memory) after surgery.

DETAILED DESCRIPTION:
Opioid-related deaths have quadrupled in the last 20 years, and nearly half of these deaths currently involve prescription opioids. Surgical patients often experience moderate-to-severe pain is common after major surgery, and surgery is associated with a 14-fold increased risk of opioid dependency compared to non-surgical controls, even after minor surgery. Furthermore, mood disorders (e.g., depression) are independently associated with persistent opioid use postoperatively, and signs of postoperative depression are common after major surgery. Thus, given these risk factors, surgical patients are at particularly high risk for opioid dependency postoperatively. Interventions that (1) reduce opioid burden, and (2) improve mood and neuropsychological function may mitigate the risk of postoperative opioid dependency. Preliminary laboratory and clinical findings demonstrate that caffeine may reduce pain after surgery, which may translate to lower opioid requirements. The study tests the hypothesis that intraoperative caffeine administration will improve opioid consumption, pain, and neuropsychological recovery in patients undergoing surgery. Through validated assessment measures, the research team will study the effects of caffeine in relation to postoperative opioid requirements, pain, and neuropsychological (e.g., cognition, depression, anxiety) trajectory after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>/= 18 years old) undergoing non-cardiac, non-neurologic, non-major vascular surgery requiring general anesthesia

Exclusion Criteria:

* Emergency surgery
* Cognitive impairment precluding capacity for informed consent
* Uncontrolled cardiac arrhythmias
* Seizure disorders
* Preoperative opioid use
* Diabetes
* Liver failure
* Pregnancy
* Breastfeeding
* Severe visual or auditory impairment (may hinder cognitive function testing)
* Patients unable to speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Vlisides, MD, Principal Investigator — Assistant Professor of Anesthesiology
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Estimate of the global volume of surgery in 2012: an assessment supporting improved health outcomes. Lancet. 2015 Apr 27;385 Suppl 2:S11. doi: 10.1016/S0140-6736(15)60806-6. Epub 2015 Apr 26. PMID 26313057
- [Background] Kundermann B, Krieg JC, Schreiber W, Lautenbacher S. The effect of sleep deprivation on pain. Pain Res Manag. 2004 Spring;9(1):25-32. doi: 10.1155/2004/949187. PMID 15007400
- [Background] Vaurio LE, Sands LP, Wang Y, Mullen EA, Leung JM. Postoperative delirium: the importance of pain and pain management. Anesth Analg. 2006 Apr;102(4):1267-73. doi: 10.1213/01.ane.0000199156.59226.af. PMID 16551935
- [Background] Lynch EP, Lazor MA, Gellis JE, Orav J, Goldman L, Marcantonio ER. The impact of postoperative pain on the development of postoperative delirium. Anesth Analg. 1998 Apr;86(4):781-5. doi: 10.1097/00000539-199804000-00019. PMID 9539601
- [Background] Karp JF, Reynolds CF 3rd, Butters MA, Dew MA, Mazumdar S, Begley AE, Lenze E, Weiner DK. The relationship between pain and mental flexibility in older adult pain clinic patients. Pain Med. 2006 Sep-Oct;7(5):444-52. doi: 10.1111/j.1526-4637.2006.00212.x. PMID 17014605
- [Background] Dolan R, Huh J, Tiwari N, Sproat T, Camilleri-Brennan J. A prospective analysis of sleep deprivation and disturbance in surgical patients. Ann Med Surg (Lond). 2016 Jan 6;6:1-5. doi: 10.1016/j.amsu.2015.12.046. eCollection 2016 Mar. PMID 26909151
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Avidan MS, Maybrier HR, Abdallah AB, Jacobsohn E, Vlisides PE, Pryor KO, Veselis RA, Grocott HP, Emmert DA, Rogers EM, Downey RJ, Yulico H, Noh GJ, Lee YH, Waszynski CM, Arya VK, Pagel PS, Hudetz JA, Muench MR, Fritz BA, Waberski W, Inouye SK, Mashour GA; PODCAST Research Group. Intraoperative ketamine for prevention of postoperative delirium or pain after major surgery in older adults: an international, multicentre, double-blind, randomised clinical trial. Lancet. 2017 Jul 15;390(10091):267-275. doi: 10.1016/S0140-6736(17)31467-8. Epub 2017 May 30. PMID 28576285
- [Background] Pandharipande P, Cotton BA, Shintani A, Thompson J, Pun BT, Morris JA Jr, Dittus R, Ely EW. Prevalence and risk factors for development of delirium in surgical and trauma intensive care unit patients. J Trauma. 2008 Jul;65(1):34-41. doi: 10.1097/TA.0b013e31814b2c4d. PMID 18580517
- [Background] Robinson TN, Raeburn CD, Tran ZV, Angles EM, Brenner LA, Moss M. Postoperative delirium in the elderly: risk factors and outcomes. Ann Surg. 2009 Jan;249(1):173-8. doi: 10.1097/SLA.0b013e31818e4776. PMID 19106695
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Nelson AM, Battersby AS, Baghdoyan HA, Lydic R. Opioid-induced decreases in rat brain adenosine levels are reversed by inhibiting adenosine deaminase. Anesthesiology. 2009 Dec;111(6):1327-33. doi: 10.1097/ALN.0b013e3181bdf894. PMID 19934879
- [Background] Gauthier EA, Guzick SE, Brummett CM, Baghdoyan HA, Lydic R. Buprenorphine disrupts sleep and decreases adenosine concentrations in sleep-regulating brain regions of Sprague Dawley rat. Anesthesiology. 2011 Oct;115(4):743-53. doi: 10.1097/ALN.0b013e31822e9f85. PMID 21857500
- [Background] Osman NI, Baghdoyan HA, Lydic R. Morphine inhibits acetylcholine release in rat prefrontal cortex when delivered systemically or by microdialysis to basal forebrain. Anesthesiology. 2005 Oct;103(4):779-87. doi: 10.1097/00000542-200510000-00016. PMID 16192770
- [Background] Pisani MA, Murphy TE, Araujo KL, Slattum P, Van Ness PH, Inouye SK. Benzodiazepine and opioid use and the duration of intensive care unit delirium in an older population. Crit Care Med. 2009 Jan;37(1):177-83. doi: 10.1097/CCM.0b013e318192fcf9. PMID 19050611
- [Background] Litaker D, Locala J, Franco K, Bronson DL, Tannous Z. Preoperative risk factors for postoperative delirium. Gen Hosp Psychiatry. 2001 Mar-Apr;23(2):84-9. doi: 10.1016/s0163-8343(01)00117-7. PMID 11313076
- [Background] Vlisides PE, Li D, McKinney A, Brooks J, Leis AM, Mentz G, Tsodikov A, Zierau M, Ragheb J, Clauw DJ, Avidan MS, Vanini G, Mashour GA. The Effects of Intraoperative Caffeine on Postoperative Opioid Consumption and Related Outcomes After Laparoscopic Surgery: A Randomized Controlled Trial. Anesth Analg. 2021 Jul 1;133(1):233-242. doi: 10.1213/ANE.0000000000005532. PMID 33939649

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 71 subjects were consented. Data is reported for a total of 60 subjects.
Period: Overall Study
Arm/Group | Experimental | Control
Started (Started is defined as randomized (n=65). Six participants were withdrawn prior to randomization.) | 34 | 31
Received Treatment | 33 | 31
Completed | 30 | 30
Not Completed | 4 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Did not receive allocated intervention | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 9 | 7 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 13 | 15 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 28 | 29 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 30 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Opioid Consumption: Postoperative Opioid Consumption, Oral Morphine Equivalents (mg)
Description: Postoperative opioid consumption, oral morphine equivalents (mg)
Time Frame: through postoperative day 3
Measure: Median (Inter-Quartile Range); unit: oral morphine equivalents (mg)
Arm/Group | Experimental | Control
Number analyzed (Participants) | 30 | 30
oral morphine equivalents (mg) | 77 [33 to 182] | 51 [15 to 117]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Other; p = 0.092, Generalized estimating equations; Median Difference (Final Values) = 55, 95% CI 2-sided [-9 to 118] — The median difference (+55) is an estimated difference between groups - rather than the actual difference - based on the pre-specified generalized estimated equations modeling

2. Secondary Outcome: Acute Pain (Patient-reported) as Assessed by Visual Analogue Scale
Description: Visual Analogue Scale (mm, 0-100, 0 = no pain, 100 = worst pain imaginable)
Time Frame: Data gathered from postoperative day 0-3. Final results were based on all values combined over this time period, per protocol.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 40 [19 to 65] | 39 [18 to 60]
Statistical Analysis 1: Comparison: Experimental vs Control; Analysis for visual analog scale scores at rest presented; Test type: Other; p = 0.802, Mixed Models Analysis

3. Secondary Outcome: Acute Pain (Observer-reported) as Assessed by Behavioral Pain Scale
Description: Behavioral Pain Scale, on a scale ranging from 3 to 12 when 3 is no pain and 12 is maximum pain
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 3 [3 to 3] | 3 [3 to 3]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Other; p = 0.320, Mixed Models Analysis

4. Secondary Outcome: Time Until Anesthetic Emergence
Description: Time from surgical dressing on to anesthetic emergence (min)
Time Frame: Duration of time from surgical dressing completion to anesthetic emergence (min); generally expected to be between 10 and 60 minutes
Population: Data at baseline or post-operative point was not available for some participants, so data is reported only for those who had complete baseline and post-operative data.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Experimental | Control
Number analyzed (Participants) | 27 | 24
Minutes | 8 [6 to 15] | 10 [6 to 17]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Other; p = 0.670, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants With Depression as Assessed by the Hospitalized Anxiety and Depression Scale (HADS-D)
Description: Number (n) of participants with positive screens (score ≥8) using the Hospitalized Anxiety and Depression Scale (HADS-D) (n, 0-21, 0 = normal, 21 = presence of severe depression symptoms)
Time Frame: baseline through postoperative day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 28 | 27
Participants | 2 | 1
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Other; p = 0.595, Fisher Exact

6. Secondary Outcome: Number of Participants With Anxiety as Assessed by the Hospitalized Anxiety and Depression Scale (HADS-A)
Description: Number (n) of participants with positive screens (score ≥8) using the Hospitalized Anxiety and Depression Scale (HADS-A) (n, 0-21, 0 = normal, 21 = presence of severe anxiety symptoms)
Time Frame: baseline through postoperative day 3
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 28 | 27
Participants | 2 | 2
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Other; p = 0.985, Fisher Exact

7. Secondary Outcome: Cognitive Function as Assessed by Trail Making Test
Description: Trail Making Test scores (seconds, 10-300,10 = fastest reported completion, 300 = maximum time allowed for completion). The change was calculated from the value at post anesthesia minus value at baseline. Higher values are considered to be worse outcomes.
Time Frame: morning of surgery baseline compared to postanesthesia care unit. Postanesthesia care unit measurement approximately 60 minutes after end of surgery
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 17 | 11
score on a scale | 10 [2 to 25] | 16 [6 to 39]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Other; p = 0.417, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Positive Affect as Assessed by PANAS (Positive and Negative Affect Schedule)
Description: Positive Affect Score (n, 10-50, 10 = least positive affect, 50 = most positive affect) via PANAS (Positive and Negative Affect Schedule)
Time Frame: postoperative day 3
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 27 | 26
score on a scale | 35 [28 to 39] | 35 [27 to 37]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Other; p = 0.432, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Negative Affect as Assessed by PANAS (Positive and Negative Affect Schedule)
Description: Negative Affect Score (n, 10-50, 10 = least negative affect, 50 = most negative affect) via PANAS (Positive and Negative Affect Schedule)
Time Frame: postoperative day 3
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 27 | 26
score on a scale | 12 [10 to 16] | 12 [10 to 17]
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Other; p = 0.673, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Percentage of Delirious Patients Per Group
Description: Number (n) of participants who has experienced at least one episode of delirium by the postoperative day 3 time point, as determined by daily Confusion Assessment Method (CAM).
Time Frame: By afternoon of postoperative day (POD) 3
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 30 | 30
Participants | 7 | 14
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Other; p = 0.058, Chi-squared

11. Other Pre Specified Outcome: Caffeine Intake: Number of Caffeinated Beverages (n) Consumed
Description: Number of caffeinated beverages (n) consumed
Time Frame: postoperative day 0-7
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Subacute Opioid Consumption: Postoperative Subacute Opioid Consumption, Oral Morphine Equivalents (mg)
Description: Postoperative subacute opioid consumption, oral morphine equivalents (mg)
Time Frame: postoperative days 4-7
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Sleep Disturbances: Incidence (%) of New, Self-reported Sleep Disturbances
Description: Incidence (%) of new, self-reported sleep disturbances
Time Frame: postoperative days 0-3
Reporting Status: Not Posted

14. Other Pre Specified Outcome: EEG Spectral Power: Spectral Power (dB) Measured on EEG
Description: Spectral power (dB) measured on EEG
Time Frame: time point 1: anesthetic emergence, approximate measurement 5-10 minutes after surgery end. Time point 2: postanesthesia care unit arrival, approximate measurement 20 minutes after end of surgery
Reporting Status: Not Posted

15. Other Pre Specified Outcome: EEG Connectivity: Connectivity (Weighted Phase Lag Index, wPLI) Measured on EEG
Description: Connectivity (weighted phase lag index, wPLI) measured on EEG
Time Frame: as for outcome 14
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Veterans Rand 12 Survey
Description: Comprehensive survey that reports on general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy /fatigue levels, social functioning and mental health. Specifically, a physical and mental health score are reported, with both score scales ranging from 0 (worst possible outcome) to 100 (best possible outcome).
Time Frame: 30 days after surgery
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Persistent Opioid Use
Description: Incidence of continued opioid use (%) on postoperative day (POD) 30
Time Frame: Postoperative day (POD) 30
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Quality of Recovery Survey
Description: Self-report outcome measure evaluating recovery after surgery and anesthesia. Scoring ranges from 3-18, 3=poor 18=excellent
Time Frame: Postoperative day (POD) 1
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Richards Campbell Sleep Questionnaire (RCSQ)
Description: Self-report instrument for measuring sleep quality. Visual Analogue Scale (mm, 0-100, 0 =Deep sleep , 100 =Light sleep)
Time Frame: Preoperative (once before surgery on day of surgery)
Population: Richards Campbell Sleep Questionnaire (RCSQ)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 58 (26) | 56 (28)

ADVERSE EVENTS:
Time Frame: Data were collected at 30 days.
Description: AEs are presented for all 64 participants who received the study drug (caffeine or placebo).
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 2/33 | 4/31
Other Adverse Events (participants affected / at risk) | 8/33 | 6/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=33) | Control (N=31)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Ileus requiring re-admittance to hospital (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Pelvic absess (Infections and infestations) | 1 (1) | 0 (0)
Hypoxia (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=33) | Control (N=31)
Ileus (Gastrointestinal disorders) | 5 (5) | 0 (0)
Nausea (General disorders) | 3 (3) | 0 (0)
Nausea with emesis (General disorders) | 0 (0) | 4 (4)
Dehydration (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT03577730/Prot_SAP_000.pdf